CLINICAL TRIAL: NCT00708890
Title: Twelve Step Based Self-help Groups for Substance Related Disorders - A Randomized Controlled Trial on a Detoxification Center
Brief Title: Twelve Step Based Self-help Groups for Substance Related Disorders
Acronym: TSF_Norway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSHF_815357
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2014-04

CONDITIONS: Substance Use Disorders
Keywords: Substance use disorders; Self-help groups; Twelve Step groups
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Brief motivation to participate in TSG
- Control group (No Intervention): Will only get a standard information about TSG group (information about meeting etc.)

INTERVENTIONS:
Behavioral: Brief motivation to participate in TSG — The intensive intervention will consist of a boost motivational session on follow-up alternatives and particularly on attending TSGs. Efforts will be made to connect the patients with TSG volunteers via the AA/NA contact telephone. The patients are encouraged to invite AA/NA contact persons to visit them on the ward. The patient will then have the possibility to be followed to a meeting after treatment. The patients in the intensive referral group will get a phone call four weeks after discharge. The focus of this call will be on continued motivation to attend TSGs.
  Arms: Intervention group

SUMMARY:
The Twelve Step groups are the most available and widespread self-help groups for patients with alcohol or drug related disorders. In a public health perspective, self-help groups (SHGs) may be considered as a supplement to professional treatment and provide aftercare soon as professional treatment has ended.

There is a need to investigate if U.S. findings and procedures concerning referrals from the health services to Twelve Step Groups (TSGs) can be replicated and accommodated to a cultural setting which is unfamiliar with these groups. There is also a particular need in the Norwegian treatment system to develop alternative treatment strategies for patients undergoing detoxification to improve their chances of long-term recovery, due to deficient formal follow-up alternatives.

We plan to carry out a RCT-study. One hundred and sixty patients entering a detoxification treatment center (Addiction Unit, Sørlandet Hospital, Kristiansand, Norway) will be assigned to two different groups: One given standard information about TSGs (brief advice) and one given intensive referral (motivational sessions and contact with TSG volunteers). A follow up assessment is planned at 6 months to determine whether intensive referral results in more TSG attendance, and if this mediates less substance use and better functioning outcomes.

This study introduces a new concept in the Norwegian health care system and relies on a systematic cooperation with user organizations (SHGs) and user volunteers. Thus the study focuses strongly on user resources.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alcohol and substance use disorders treated on a detox ward

Exclusion Criteria:

* Severe psychiatric comorbidity
* Patients on opioid replacement therapy
* Those who have appointment with other inpatient treatment at intake (and will be transferred to such treatment)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Self-help groups attendance and involvement during 6 months observation period. | Six months after detox treatment

SECONDARY OUTCOMES:
1)Substance use outcomes measured by Europ-ASI 2) Quality of Life | 6 months after detox treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sørlandet Sykehus, Kristiansand, VA, Norway

REFERENCES:
- [Result] Vederhus JK, Timko C, Kristensen O, Clausen T. The courage to change: patient perceptions of 12-Step fellowships. BMC Health Serv Res. 2011 Dec 15;11:339. doi: 10.1186/1472-6963-11-339. PMID 22171827
- [Result] Vederhus JK, Timko C, Kristensen O, Hjemdahl B, Clausen T. Motivational intervention to enhance post-detoxification 12-Step group affiliation: a randomized controlled trial. Addiction. 2014 May;109(5):766-73. doi: 10.1111/add.12471. Epub 2014 Feb 16. PMID 24400937
- See also: The Norwegian Centre for Addiction Research web site — http://www.seraf.uio.no/forskning/Interaktivt%20forum/Registrerte%20forskningsprosjekter/gruppe3/Vederhus.pdf